CLINICAL TRIAL: NCT00346281
Title: A Phase IIa, Safety Study of the Active Implantable(Radiological) Medical Device 32P BioSilicon, Administered Intratumourally to Patients With Advanced, Unresectable Pancreatic Cancer, in Addition to Standard IV Gemcitabine Chemotherapy
Brief Title: 32P BioSiliconTM in Addition to Gemcitabine in Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: pSiMedica Limited (Industry)
Collaborators: pSiOncology Private Limited (Unknown); Singapore General Hospital (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB2-201
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2006-06-29 (Estimated); Status verified 2006-06

CONDITIONS: Pancreatic Cancer
Keywords: unresectable pancreatic cancer; brachytherapy; 32P; BioSilicon; locally advanced; gemcitabine; intratumourally; unresectable
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Device: 32P BioSilicon

SUMMARY:
This is the first study investigating the safety of 32P BioSilicon in patients with advanced,unresectable pancreatic cancer who are also receiving standard intravenous gemcitabine chemotherapy. The secondary aims of the study will assess the implantation procedure, localisation of 32P BioSilicon, tumour response and survival parameters.

Tumours targetted with 32P BioSilicon is hypothesized to show a reduction in tumour volume and with the low radioactivity dose that is delivered intratumourally, the incidence of side effects associated with the treatment is expected to be low. Prologation of survival and improved quality of life could be favourable outcomes of the investigational product.

DETAILED DESCRIPTION:
This will be an open label, Phase IIa safety study recruiting about 15 patients from at least two sites. All patients will have 32P BioSilicon implanted into the pancreatic tumour as a single implant, using endoscopic ultrasound. The study will examine the safety of an injected activity equivalent to an absorbed dose of 100 Gy (which is considered to be an initial low risk radioactivity level), administered intratumourally to patients with pancreatic cancer. All patients will receive gemcitabine treatment within 2 weeks prior to or within 3 days of implantation. Any dose adjustments to the gemcitabine treatment will be made according to the clinical judgement of the oncologist in the team and this will be made in accordance with the current approved prescribing receommendations. Implantation of 32P BioSilicon will be performed endoscopically by a trained endoscopist and a nuclear medicine physician. The 32P BioSilicon will be prepared by a designated personnel licenced to handle radioactive products and all radioactive waste will be handled and managed as per the institution's guidelines and in compliance with local regulatory requirements. Bremsstrahlung imaging will be performed post implantation as a preliminary indication of localisation of the implanted 32P BioSiliconTM.

Assessments will be performed for haematology, biochemistry, CA19-9 marker, performance status and any adverse event observed or reported will be graded according to the CTCAE. To minimise inter-observer variation, the patient should be assessed by the same investigator throughout the study. Tumour assessment and tumour volume calculation will be performed by designated radiologists who are independent of the study. To standardise, the CT scans will be performed according to an agreed scanning protocol and the images will be captured in a DICOM format at site for assessment by the independent radiologist. Tumour response will be evaluated only for target tumours using RECIST.

Pain assessment using the Brief Pain Inventory (BPI) pain score will be recorded by the patient.

Patients who have clinically and/or radiologically stable or responding disease have the option to continue gemcitabine, at the discretion of the investigator. Following discontinuation from the study, patients will be followed up for progression-free, and overall survival.

A Data Monitoring Committee will review the study data at regular teleconference throughout the study.

ELIGIBILITY:
Inclusion Criteria: -

* Histologically proven locally advanced or metastatic adenocarcinoma of the pancreas
* Advanced pancreatic disease, not amenable to surgical resection
* Measurable disease by CT scan, with a tumour burden equivalent to a diameter of no less than 3cm and no greater than 6cm
* ECOG Performance status 0 - 2
* Life expectancy at least three months
* Laboratory parameters:

Hb greater than or equal to 10 g/dl Platelets greater than or equal to 100,000 mm3 ANC greater than or equal to 1500/mm3 Bilirubin < 1.3 x ULN Alkaline phosphatase < 5 x ULN Transaminases < 5 x ULN Creatinine < 1.5 x ULN Prothrombin (PT) and partial thromboplastin time (PTT) within normal range Serum calcium within normal range

* All patients of reproductive potential must agree to use an effective barrier method of contraception during the study and for six months following termination of treatment.
* Male and female patients aged 18 or over who have provided written informed consent

Exclusion Criteria: -

* Any previous treatment with 32 Phosphorus or with 32P BioSiliconTM
* Any prior radiotherapy for pancreatic cancer
* Use of other investigational agent at the time of enrolment, or within 30 days or five half-lives of enrolment, whichever is longer
* History of hypersensitivity to any of the study products or to products with similar chemical structures (i.e. silicon or phosphorous)
* History of malignancy of any other organ system, treated or untreated, within the past five years whether or not there is evidence of local recurrence or metastases, with the exception of localised basal cell carcinoma of the skin and in situ cervical carcinoma
* Pregnant or lactating women
* Significant tumour related pain for which analgesic intervention incorporating epidural or EUS is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-06; Study Completion 2008-06

PRIMARY OUTCOMES:
Safety profile of the patients defined by the Adverse Events profile.

SECONDARY OUTCOMES:
Will assess ease of use, tumour response, duration of response, progression free survival and overall survival. Target tumour response summaries for the study will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce KH Chow, MBBS, PhD, Principal Investigator — Singapore General Hospital; Paul Ross, MBBS,PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (2):
- Singapore General Hospital, Outram Road, Singapore
- Guy's and St Thomas' Hospital NHS Trust, London, United Kingdom

REFERENCES:
- See also: BrachySil A Novel Targeted Cancer Therapy — http://www.psivida.com